CLINICAL TRIAL: NCT06089980
Title: Observing the Acute Effects Following a Single Oral Dose of Kratom and Effects Following Kratom Cessation Among Adults Who Use Regularly.
Brief Title: Direct Observation Study of Kratom Product Effects Among Regular Consumers
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Florida (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00408134; R00DA055571 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Kratom Pharmacokinetics; Kratom Pharmacodynamics; Kratom
Keywords: kratom

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human urine; plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute kratom exposure: Participants who regularly consume kratom will orally self-administer a single serving of the participants commercial kratom product under direct observation in order to evaluate acute physiological, subjective, and cognitive effects and determine pharmacokinetics. This will occur during the first 24 hours of study participation. Participants will undergo direct observation and assessment for after ceasing all kratom product use. Physiological, subjective, and cognitive effects during this supervised withdrawal will be assessed.
  Interventions: Behavioral: Effects from acute kratom exposure

INTERVENTIONS:
Behavioral: Effects from acute kratom exposure — Participants who regularly use commercial Kratom products will orally consume a known quantity of kratom under direct observation on first study day; following this, participants will stop kratom use for approximately 2 nights and 2.5 days for the duration of the study.

SUMMARY:
The goal of this observational clinical study is to is to learn more about how commercial kratom products affect healthy adults who consume them regularly. The main questions it aims to answer are:

1. What are the acute physiological, subjective, and cognitive effects of kratom following participant self-administration of a single oral dose of the participants usual kratom product at the participants typical dose?
2. What are the physiological, subjective, and cognitive effects associated with kratom product discontinuation among adults who use regularly?
3. What are the pharmacokinetics of kratom products consumed by adults who use regularly? On the first study day: Under direct observation, participants will self-administer a single oral dose of the participants own commercial kratom product that that is regularly taken and will consume it at the participants self-selected typical dose/serving. Following this, serial blood draws and urine collection will occur along with administration of validated questionnaires, tests, and continual monitoring. After this first study day, participants will no longer be permitted to use any of the participants kratom product during the study. On study nights/days 2-3: participants will reside a clinical research unit and be observed and evaluated for kratom withdrawal syndrome.

ELIGIBILITY:
INCLUSION CRITERIA:

1. >21 years
2. reporting kratom use >5 times per week for >3 months prior to study screening
3. English language proficiency
4. Willingness to provide requested samples of the kratom product being currently taken

EXCLUSION CRITERIA:

1. Reports any acute adverse, unexpected, or otherwise sudden health event related to the typical kratom product dose that occurred within 30 days of screening
2. Having ever sought medical attention for an acute adverse health event as a result of taking any kratom product.
3. Cannot or will not provide kratom product samples in the form of an unopened package of kratom that is clearly labeled with at least the product and vendor name.
4. Self-reports using kratom products by any other route than orally swallowing.
5. Current physical dependence on alcohol, benzodiazepines, or opioids
6. Reports use of fentanyl within the past month and/or has a fentanyl positive drug screen.
7. Discordance between self-reported substance use and drug screen results obtained during screening.
8. Lifetime or current psychotic disorder
9. Current untreated major depressive or bipolar disorder
10. Pregnancy or nursing
11. Physical, psychiatric, or environmental conditions considered by study team to increase risk or undue burden (e.g., untreated hypertension, high BMI, etc.).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 21 or older who use kratom.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Peak subjective opioid withdrawal score | Up to 3 days
  Peak score on the Subjective Opioid Withdrawal Scale (SOWS); that occurs between Study Days 1-3. Score range 0-64. 5-point scale of intensity: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely. Higher score indicates higher intensity. SOWS will be administered at 8 time points on Study Days 1-2 and 7 time points on Study Day 3.
Time in minutes until a Subjective Opioid Withdrawal (SOWS) score of more than 11 is reached | up to 3 days
  Time, in minutes, until at least a moderate score (of 11 or higher) is reached on the Subjective Opioid Withdrawal Scale (SOWS). SOWS will be administered at 8 time points on Study Days 1-2 and 7 time points on Study Day 3. 5-point scale of intensity: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely. Score range 0-64. Higher score indicates higher intensity.
Peak rating and changes in rating on Drug Effects Questionnaire (primary subjective outcome) | Up to 3 days
  Drug Effects Questionnaire (DEQ) visual analogue scale (0-100) rating for DEQ item "feeling high." The DEQ will be administered at 7 timepoints on Study Day 1 and at 6 times points on Study Days 2 and 3.
Peak rating and change in rating on Drug Effects Questionnaire (primary subjective outcome) | Up to 3 days
  Drug Effects Questionnaire (DEQ) visual analogue scale (0-100) rating for DEQ item "drug liking." The DEQ will be administered at 7 time points on Study Day 1 and at 6 times points on Study Days 2 and 3.
Changes in accuracy on psychomotor task (primary cognitive outcome) | Up to 3 days
  The 2-minute computerized Digit Symbol Substitution Task (DSST) outcome of total number of correct responses (accuracy) within the 2-minute test window. This will evaluate cognitive performance and impairment. The DSST will be administered at 7 time points on Study Day 1 and at 6 times points on Study Days 2 and 3.
Pupil diameter nadir size as measured in millimeters (mm) (primary physiological outcome). | Up to 3 days
  Pupil diameter in mm under stable light conditions using a pupilometer. Pupil size will be measured at 8 timepoints on Study Days 1 and 2 and at 7 timepoints on Study Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Smith, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No